CLINICAL TRIAL: NCT00002899
Title: Phase III Trial on Convergent Beam Irradiation of Cerebral Metastases
Brief Title: Adjuvant Radiation Therapy in Treating Patients With Brain Metastases
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22952-26001; EORTC-22952; EORTC-26001
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy; Radiosurgery

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Adjuvant radiation therapy may kill any remaining tumor cells following surgery or radiosurgery for brain metastases.

PURPOSE: This randomized phase III trial is studying surgery or radiosurgery alone to see how well it works compared to surgery or radiosurgery and whole-brain radiation therapy in treating brain metastases in patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Investigate the efficacy and toxicity of adjuvant whole brain radiotherapy after prior surgical resection or radiosurgery of 1 to 3 brain metastases from solid tumor in patients with good performance status and controlled systemic cancer.

Secondary

* Determine overall survival and progression-free survival of patients treated on this protocol.
* Determine time to neurologic progression in patients treated on this protocol.
* Determine quality of life of patients treated on this protocol.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating center, number of brain metastases (single vs multiple), type of primary tumor (stable systemic cancer vs synchronous or unknown primary), WHO performance status (0-1 vs 2), and treatment (prior surgical resection vs planned radiosurgery).

Patients who have undergone complete surgical resection are randomized to 1 of 2 treatment arms within 4 weeks after surgery.

* Arm I: Patients undergo adjuvant whole brain radiotherapy (WBRT).
* Arm II: Patients do not receive adjuvant radiotherapy. Patients planning to undergo radiosurgery are randomized to 1 of 2 treatment arms.
* Arm III: Patients undergo radiosurgery followed by adjuvant WBRT within 4 weeks after surgery.
* Arm IV: Patients undergo radiosurgery alone. Quality of life is assessed at baseline, at 8 weeks, and then every 3 months thereafter.

After completion if study treatment, patients are followed at 8 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 340 patients (85 per treatment arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of brain metastases from a histologically confirmed primary or metastatic extracranial tumor, meeting 1 of the following criteria:

  * Stable systemic cancer for the last 3 months (achieved by surgery, radiotherapy, chemotherapy, or hormonal therapy), defined as absence of symptomatic or radiological progression
  * Asymptomatic synchronous primary tumor (treatable by surgery, radiotherapy, chemotherapy, or hormonal therapy)

    * No metastases outside the CNS
  * Unknown primary tumor
* Must have one to three brain lesions, confirmed by enhanced MRI prior to radiosurgery or surgery

  * No brain stem metastases
  * No leptomeningeal metastases
  * No brain metastases from small cell lung cancer, lymphoma, leukemia, myeloma, or germ cell tumors
* Patients planning to undergo radiosurgery must meet the following criteria:

  * Largest diameter ≤ 3.5 cm for single metastasis
  * Largest diameter ≤ 2.5 cm for multiple metastases
  * Stereotactic biopsy required if not extracranial tumor (unknown primary tumor) OR extracranial diagnosis made more than 4 years previously
* Prior neurosurgery patients must have undergone complete surgical resection
* No recurrent brain metastases after prior surgery and/or radiosurgery and/or brain radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2 (may be assessed under steroid therapy)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No concurrent chemotherapy during whole brain radiotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 1996-11; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Survival with a WHO performance status 0-2 as measured by Logrank at 8 weeks after completion of study treatment, and then every 3 months until death

SECONDARY OUTCOMES:
Overall survival as measured by Logrank at 8 weeks after completion of study treatment, and then every 3 months until death
Progression-free survival as measured by Logrank 8 weeks after completion of study treatment, and then every 3 months until death
Time to neurological progression as measured by Logrank 8 weeks after completion of study treatment, and then every 3 months until death
Acute toxicity as measured by EORTC and RTOG scale 8 weeks after completion of study treatment, and then every 3 months until death
Late toxicity as measured by Subjective, Objective, Management and Analytic/Late Effects on Normal Tissues (SOMA/LENT) scale 8 weeks after completion of study treatment, and then every 3 months until death
Quality of life as measured by QLQ-C30 and BN-25 8 weeks after completion of study treatment, and then every 3 months until death

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Peter Mueller, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne; Riccardo Soffietti, MD, Study Chair — Universita Degli Studi di Turin
Locations (33):
- Belgium (3):
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - U.Z. Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- Helsinki University Central Hospital, Helsinki, Finland
- France (7):
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Centre Haute Energie, Nice
  - CHU Pitie-Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
- Germany (4):
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Medizinische Klinik und Poliklinik III - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Tuebingen, Tübingen
  - Heinrich-Braun-Krankenhaus Zwickau, Zwickau
- Rambam Medical Center, Haifa, Israel
- Italy (5):
  - Ospedale Niguarda Ca'Granda, Milan
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Ospedale Ostetrico Ginecologica Sant Anna, Torino
  - Universita Degli Studi di Turin, Torino
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano, Torino
- Paula Stradina Kliniskas Universitates Slimnica, Riga, Latvia
- Maastro Clinic - Locatie Maastricht, Maastricht, Netherlands
- Hospital Santa Maria, Lisbon, Portugal
- Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona, Spain
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (6):
  - University College Hospital - London, London, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Royal Preston Hospital, Preston, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Result] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Result] Mekhail T, Sombeck M, Sollaccio R. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. Curr Oncol Rep. 2011 Aug;13(4):255-8. doi: 10.1007/s11912-011-0180-1. No abstract available. PMID 21584645
- [Derived] Churilla TM, Chowdhury IH, Handorf E, Collette L, Collette S, Dong Y, Alexander BM, Kocher M, Soffietti R, Claus EB, Weiss SE. Comparison of Local Control of Brain Metastases With Stereotactic Radiosurgery vs Surgical Resection: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2019 Feb 1;5(2):243-247. doi: 10.1001/jamaoncol.2018.4610. PMID 30419088
- [Derived] Churilla TM, Handorf E, Collette S, Collette L, Dong Y, Aizer AA, Kocher M, Soffietti R, Alexander BM, Weiss SE. Whole brain radiotherapy after stereotactic radiosurgery or surgical resection among patients with one to three brain metastases and favorable prognoses: a secondary analysis of EORTC 22952-26001. Ann Oncol. 2017 Oct 1;28(10):2588-2594. doi: 10.1093/annonc/mdx332. PMID 28961826
- [Derived] Soffietti R, Kocher M, Abacioglu UM, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Mueller RP, Tridello G, Collette L, Bottomley A. A European Organisation for Research and Treatment of Cancer phase III trial of adjuvant whole-brain radiotherapy versus observation in patients with one to three brain metastases from solid tumors after surgical resection or radiosurgery: quality-of-life results. J Clin Oncol. 2013 Jan 1;31(1):65-72. doi: 10.1200/JCO.2011.41.0639. Epub 2012 Dec 3. PMID 23213105